CLINICAL TRIAL: NCT05212519
Title: Correlation of Vitamin D Levels in Early Pregnancy With Gestational Diabetes and Pregnancy Outcomes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Min Shang (Other)
Responsible Party: Sponsor-Investigator, Min Shang, Chief Physician, Department of Obstetrics and Gynecology, Beijing Friendship Hospital, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: rszqwssdspyrsqtnbjrsjjdxgx
Record Dates: First submitted 2021-12-29; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: GDM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum 25-(OH)D3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 25-hydroxyvitamin D3≥30 ng/ml: the patients were categorized as having vitamin D sufficiency if its concentrationis ≥30 ng/m
- 25-hydroxyvitamin D3< 30 ng/ml: insufficiency if levels are <30 but ≥20 ng/ml, deficiency when levels are <20 but ≥10 ng/ml and severe deficiency with levels <10 ng/ml

INTERVENTIONS:
Other:  — For observational research
  Groups: 25-hydroxyvitamin D3< 30 ng/ml

SUMMARY:
Explore the specific correlation between different concentration levels of vitamin D in early pregnancy and blood glucose levels at each time node of OGTT, the correlation between different concentrations of vitamin D levels and A1 and A2 diabetes in pregnancy, and the impact on maternal and infant outcomes , And provide a basis for the prevention and treatment of GDM.

DETAILED DESCRIPTION:
1. According to the diagnostic criteria of GDM proposed by the International Association for the Study of Diabetes and Pregnancy (IADPSG), the 18-45-year-old pregnant women who were filed and delivered by the Obstetrics Department of Beijing Friendship Hospital from September 2022 to September 2024 were selected to collect their early pregnancy (pregnancy 1- 3 months) Vitamin d level, divided into three groups: A (<20 ng/ml), B (20~<30 ng/ml), and C (≥30 ng/ml), compare the early pregnancy (1-3 months of pregnancy) Differences in vitamin D levels.
2. Follow-up patients with gestational diabetes mellitus are divided into type A1 gestational diabetes patients (GDM 1 group) and type A2 gestational diabetes patients (GDM 2 group) according to whether participant are treated with insulin, and study vitamins through multiple linear and logistic regression models The relationship between D level and GDM and follow-up pregnancy outcome
3. Analyze the relationship between the level of vitamin D in early pregnancy and pregnancy complications, such as whether it is combined with premature rupture of membranes, hypertension during pregnancy, whether it is a cesarean section, whether it is a giant baby, whether there is asphyxia in newborns, etc.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18 to 45 years who have received regular antenatal examinations and delivered in the department of obstetrics in Beijing Friendship Hospital, Capital Medical University.

Exclusion Criteria:

(1) chronic or acute disease history (diabetes mellitus, hypertension,or thyroid disease); (2) any mental disorder; (3) abortion (fetal loss before 28 gestational weeks); (4)multiple fetuses; (5) planning to give birth in other hospitals.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women aged 18 to 45 years who have received regular antenatal examinations and delivered in the department of obstetrics in Beijing Friendship Hospital, Capital Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Whether suffering from gestational diabetes | 2022-1-1to2024-1-1
  Low vitamin D levels are more likely to develop diabetes

CONTACTS AND LOCATIONS:
Overall Officials: min shang, MedicalPhD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
no plan